CLINICAL TRIAL: NCT06172543
Title: The Effects of Protein and Carbohydrate Supplementation, With and Without Creatine, on Occupational Performance in Firefighters
Brief Title: The Effects of Nutritional Supplementation on Occupational Performance in Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ward Dobbs (Other)
Collaborators: Mayo Clinic (Other); Des Moines University (Other); Lindenwood University (Other)
Responsible Party: Sponsor-Investigator, Ward Dobbs, Assistant Professor, University of Wisconsin, La Crosse
Organization: University of Wisconsin, La Crosse (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UWisconsinLaCrosse
Record Dates: First submitted 2023-11-22; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Fatigue
Keywords: Creatine
MeSH Terms: conditions — Fatigue | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine Monohydrate Group (Experimental): 25 grams of Whey Protein Isolate + 25 grams of Carbohydrate Powder + 5 grams of Creatine
  Interventions: Dietary Supplement: Creatine Monohydrate
- Non Creatine Group (Placebo Comparator): 25 grams of Whey Protein Isolate + 25 grams of Carbohydrate Powder only
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — Participants were assigned to ingest a single serving daily of either A) a 25-gram dose of whey protein isolate + 25-gram dose of carbohydrate powder (ProCarb); or B) a 25-gram dose of Whey Protein Isolate + 25-gram dose of carbohydrate powder + 5-gram dose of creatine monohydrate (Creatine) for a 17-21-day period.
  Arms: Creatine Monohydrate Group
Dietary Supplement: Control — A 25-gram dose of whey protein isolate + 25-gram dose of carbohydrate powder (ProCarb)
  Arms: Non Creatine Group

SUMMARY:
The purpose of this study was to assess the usefulness of protein and carbohydrate supplementation, with and without creatine, on occupational performance in firefighters. Research has examined the effects of adding creatine to whey protein and carbohydrates on training adaptations in resistance-trained individuals with mixed finding.

Furthermore, the ergogenic benefit of protein and carbohydrate supplementation, with or without creatine, in firefighters is largely unknown. Therefore, the primary aim of the current study was to examine the effects of protein and carbohydrate supplementation, with or without creatine, on occupational performance in firefighters.

ELIGIBILITY:
Inclusion Criteria:

* Being a firefighter between the ages of 18-55 years of age, and medically cleared for field duty.

Exclusion Criteria:

* Any current musculoskeletal or neurological condition that would prohibit the completion of performance testing.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Time to completion | 24 Days
  Time to completion for tasks including a hose carry, body drag, stair climb, and forcible entry (Keiser sled hammer) for time. For the hose carry, firefighters advanced a 30.48 m section of a charged 4.45 cm hose line over a distance of 30.5 m in a straight line before flowing water for 2 seconds. Rescue consisted of firefighters being instructed to grasp a mannequin (mass 50 kg, height: 180 cm) underneath the shoulders using a "seatbelt" grip and dragging the mannequin 30.5 m backward. This test is known as the body drag. Stair climb consisted of climbing four flights of stairs and returning to the bottom as quickly as possible. In the forcible entry, firefighters struck a simulated forcible entry chopping device (Keiser FORCE Machine, Keiser Co., USA) using a 3.6 kg sledgehammer until completed. The total time to complete each task was recorded, in addition to the total completion time for all tasks summed together.
Time Trial | 24 Days
  A maximal effort, 3.5 km time trial on an air-braked cycle ergometer (Assault Bike, As-sault Fitness Products, Carlsbad, CA, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Jagim, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Fire Department, La Crosse, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data is available upon request.